CLINICAL TRIAL: NCT01485172
Title: A Fixed Dose, Dose Response Study for Ropinirole Prolonged Release (PR) in Patients With Early Stage Parkinson's Disease
Brief Title: A Fixed Dose, Dose Response Study for Ropinirole Prolonged Release in Patients With Early Stage Parkinson's Disease
Acronym: TANDEM-662
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 111662
Record Dates: First submitted 2011-12-01; First posted 2011-12-05 (Estimated); Results first posted 2015-02-02 (Estimated); Last update posted 2018-06-20 (Actual); Status verified 2018-06

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ropinirole (Experimental): ropinirole 2, 4, 8, 12, or 24 mg/day
  Interventions: Drug: ropinirole monotherapy
- placebo (Placebo Comparator): placebo comparator 2, 4, 8, 12, or 24 mg/day
  Interventions: Drug: ropinirole monotherapy; Drug: placebo monotherapy

INTERVENTIONS:
Drug: ropinirole monotherapy — ropinirole as monotherapy in Parkinson's disease
Drug: placebo monotherapy — placebo as monotherapy in Parkinson's disease
  Arms: placebo

SUMMARY:
This study is a fixed dose, dose response study to characterize the dose response for ropinirole PR in early stage PD patients (Hoehn & Yahr stages I-III). After screening and baseline assessments, subjects will be randomized to one of six final target treatment groups (placebo, 2, 4, 8, 12 or 24mg/day ropinirole PR). The study will consist of a screening period, an up-titration period, a maintenance period, a down titration period and a follow up period. This study utilizes change from baseline in the UPDRS motor score as the primary endpoint, in line with that used in the ropinirole PR monotherapy pivotal study (SK&F101468/168). Clinical review of the primary and secondary endpoints will be performed in order to establish the lowest maximally effective therapeutic dose.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic Parkinson's disease (according to modified Hoehn & Yahr criteria Stages I-III.)
* Subjects aged 30 years or greater at screening. Women of child-bearing potential must be practicing a clinically accepted method of contraception during the study and for at least one month prior to randomization and one month following completion of the study. Acceptable contraceptive methods include abstinence, oral contraception, injectable progestogen, implants of levonorgestrel, estrogenic vaginal ring, percutaneous contraceptive patches, surgical sterilisation, male partner sterilization, intrauterine device [IUD], or double barrier method: condom or occlusive cap (diaphragm or cervical/vault caps) plus spermicidal agent (foam/gel/film/cream/suppository.
* A baseline UPDRS motor score of at least 10.
* Limited prior exposure to low or moderate doses of L-DOPA (up to 3 months in total) or dopamine agonists including ropinirole (up to 6 months in total) is allowed provided treatment is discontinued for a minimum of 4 weeks prior to screening.
* Provide written informed consent for this study.
* Be willing and able to comply with study procedures.

Exclusion Criteria:

* Subjects with Parkinson's disease in whom dopaminergic therapy is not warranted at the time of screening.
* Subjects with severe, clinically significant condition(s) other than Parkinson's disease which, in the opinion of the investigator, render the subject unsuitable for the study (e.g., psychiatric, haematological, renal, hepatic, endocrinology, neurological [other than Parkinson's disease], cardiovascular, or active malignancy [other than basal cell carcinoma]).
* Subjects with crippling degenerative arthritis or other physical or mental conditions precluding accurate assessment of efficacy or safety.
* Subjects with prior or current major psychosis (e.g., schizophrenia or psychotic depression) e.g. scoring 3 or 4 on UPDRS item 2 [thought disorder] or item 3 [depression].
* Subjects with severe clinical dementia e.g. scoring 3 or 4 on UPDRS item 1 [mentation].
* Subjects with severe dizziness or fainting due to postural hypotension on standing.
* Subjects with a personal history of melanoma.
* Subjects with clinically significant abnormalities in laboratory or ECG tests at Screening. If findings are outside the normal range and the subject is included, it must be documented by the investigator that the findings are not of clinical significance.
* Subjects diagnosed with an impulse control disorder. The modified MIDI will be conducted at screening. Subjects who score positive for this screen must be referred to a specialist for diagnostic evaluation prior to enrolling (screening) in the study.
* Subjects with an active suicidal plan/intent or have had active suicidal thoughts in the past 6 months. Subjects with a history of suicide attempt in the last 2 years or more than 1 lifetime suicide attempt.
* Current alcohol or drug dependence.
* Definite or suspected personal or family history of clinically significant adverse reactions or hypersensitivity to ropinirole (or to drugs with a similar chemical structure) that would preclude long-term dosing with ropinirole.
* Withdrawal, introduction, or change in dose of hormone replacement therapy and/or any drug known to substantially inhibit CYP1A2 (e.g. ciprofloxacine, fluvoxamine, cimetidine, ethinyloestradiol) or induce CYP1A2 (e.g. tobacco, omeprazole) within 7 days prior to baseline (randomization).
* Subjects on chronic therapy with any of these agents may be enrolled but doses must have remained stable from 7 days prior to baseline (randomization) through the end of the treatment period. Smokers should maintain normal smoking habit.
* Women who are pregnant or breast-feeding.
* Use of an investigational drug from 30 days or 5 half-lives (which ever is longer) prior to baseline (randomization) to the end of the treatment period.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2012-01-31 (Actual); Primary Completion 2014-04-30 (Actual); Study Completion 2014-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (31):
- United States (11):
  - GSK Investigational Site, Fountain Valley, California
  - GSK Investigational Site, Pasadena, California
  - GSK Investigational Site, Reseda, California
  - GSK Investigational Site, Torrance, California
  - GSK Investigational Site, Ventura, California
  - GSK Investigational Site, Boca Raton, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Augusta, Georgia
  - GSK Investigational Site, Forest Hills, New York
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Richmond, Virginia
- Estonia (2):
  - GSK Investigational Site, Tallinn
  - GSK Investigational Site, Tartu
- Russia (12):
  - GSK Investigational Site, Chelyabinsk
  - GSK Investigational Site, Kazan'
  - GSK Investigational Site, Krasnoyarsk
  - GSK Investigational Site, Kursk
  - GSK Investigational Site, Novosibirsk
  - GSK Investigational Site, Omsk
  - GSK Investigational Site, Perm
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Saratov
  - GSK Investigational Site, Smolensk
  - GSK Investigational Site, Ufa
  - GSK Investigational Site, Yekaterinburg
- Slovakia (2):
  - GSK Investigational Site, Banská Bystrica
  - GSK Investigational Site, Bratislava
- South Korea (4):
  - GSK Investigational Site, Busan
  - GSK Investigational Site, Donggu Gwangju
  - GSK Investigational Site, Seoul
  - GSK Investigational Site, Sungnam -Gyeonggi-do

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 111662 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 111662 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 111662 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 111662 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 111662 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 111662 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible participants (par.) were diagnosed with early stage Parkinson's disease (according to modified Hoehn and Yahr criteria Stages I-III) and randomized at Screening into one of six treatment arms to receive placebo or ropinirole Prolonged Release (PR) tablets.
Pre-assignment Details: After Screening, par. underwent a 13 Week Up-Titration Period until reaching their target dose then continued on their target dose during a 4 Week Maintenance Period up to Week 17. All par. underwent a 1 Week Down-Titration Period and then a Follow-Up Visit 1-2 Weeks after receiving the last dose of treatment.
Groups:
- Treatment Group A: Placebo: Participants (par.) were administered a matching Prolonged Release (PR) placebo tablet Once Daily (OD) for up to 17 weeks. Par. completed a Follow-up visit 2 weeks after receiving the last dose of study medication.
- Treatment Group B: 2 mg/Day: Par. were administered a ropinirole PR tablet totalling 2 milligrams per day (mg/day), OD up to Study Week 17. Par. reaching their target dose and completing the maintenance period or withdrawing prematurely were switched to placebo for down-titration for 1 week before completing a Follow-up visit 2 weeks after receiving the last dose of study medication.
- Treatment Group C: 4 mg/Day: Par. were administered a ropinirole PR tablet totalling 2 mg/day, OD for one week. Par. were up-titrated to 4 mg/day at Week 2 and continued this dose up to Study Week 17. Par. reaching their target dose and completing the maintenance period or withdrawing prematurely were down-titrated to 2 mg for 4 days and then switched to placebo for 3 days for down-titration before completing a Follow-up visit 2 weeks after receiving the last dose of study medication.
- Treatment Group D: 8 mg/Day: Par. were administered a ropinirole PR tablet totalling 2 mg/day, OD for one week. Par. were up-titrated to 4 mg/day at Week 2, 6 mg/day at Week 3, and 8 mg/day at Week 4. Par. continued this dose up to Study Week 17. Par. reaching their target dose and completing the maintenance period or withdrawing prematurely were down-titrated for 1 week before completing a Follow-up visit 2 weeks after receiving the last dose of study medication.
- Treatment Group E: 12 mg/Day: Par. were administered a ropinirole PR tablet totalling 2 mg/day, OD for one week. Par. were up-titrated to 4 mg/day at Week 2, 6 mg/day at Week 3, 8 mg/day at Week 4, and 12 mg/day at Week 6. Par. continued this dose up to Study Week 17. Par. reaching their target dose and completing the maintenance period or withdrawing prematurely were down-titrated for 1 week before completing a Follow-up visit 2 weeks after receiving the last dose of study medication.
- Treatment Group F: 24 mg/Day: Par. were administered a ropinirole PR tablet totalling 2 mg/day, OD for one week. Par. were up-titrated to 4 mg/day at Week 2, 6 mg/day at Week 3, 8 mg/day at Week 4, 12 mg/day at Week 6, 16 mg/day at Week 8, 20 mg/day at Week 10, and 24 mg/day at Week 12. Par. continued this dose up to Study Week 17. Par. reaching their target dose and completing the maintenance or withdrawing prematurely were down-titrated for 1 week before completing a Follow-up visit 2 weeks after receiving the last dose of study medication.
Period: Overall Study
Arm/Group | Treatment Group A: Placebo | Treatment Group B: 2 mg/Day | Treatment Group C: 4 mg/Day | Treatment Group D: 8 mg/Day | Treatment Group E: 12 mg/Day | Treatment Group F: 24 mg/Day
Started | 40 | 13 | 41 | 40 | 39 | 13
Completed | 33 | 12 | 34 | 32 | 34 | 9
Not Completed | 7 | 1 | 7 | 8 | 5 | 4
Not completed — Adverse Event | 2 | 1 | 2 | 2 | 1 | 2
Not completed — Lack of Efficacy | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 4 | 5 | 1 | 0
Not completed — Protocol defined stopping criteria | 1 | 0 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Group A: Placebo | Treatment Group B: 2 mg/Day | Treatment Group C: 4 mg/Day | Treatment Group D: 8 mg/Day | Treatment Group E: 12 mg/Day | Treatment Group F: 24 mg/Day | Total
Number analyzed (Participants) | 40 | 13 | 41 | 40 | 39 | 13 | 186
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.1 (8.82) | 58.2 (11.12) | 62.1 (11.38) | 60.3 (11.72) | 61.7 (10.78) | 62.5 (12.88) | 61.6 (10.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 5 | 16 | 28 | 19 | 6 | 91
  Male | 23 | 8 | 25 | 12 | 20 | 7 | 95
Race/Ethnicity, Customized [Number; unit: Participants]
  African American/African Heritage | 2 | 0 | 0 | 0 | 0 | 0 | 2
  Asian - East Asian | 2 | 0 | 1 | 5 | 2 | 1 | 11
  Asian - Japanese | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Asian - South East Asian Heritage | 0 | 0 | 0 | 1 | 0 | 0 | 1
  White - White/Caucasian | 36 | 13 | 39 | 34 | 36 | 12 | 170
  Missing | 0 | 0 | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline (BL) in Unified Parkinson Disease (PD) Rating Scale (UPDRS) Motor Score
Description: The UPDRS is a clinician based rating scale used to measure motor impairments and disability. The UPDRS assesses six features of PD impairment. These are evaluated using a combination of data collected by interview and examination of the participant. One of the six features include the Part III - Motor Examination where scores can range 0-108 where the maximum score indicates the worse condition. BL is defined as the last non-missing assessment measured on or before the first dose date. The change from BL was calculated by subtracting the BL values from the individual post-randomization values. The least squares(LS) means were estimated using the mixed model repeated measures(MMRM) adjusting for BL UPDRS motor score and race(white versus other) or by using the non-parametric rank analysis of covariance(ANCOVA).
Time Frame: Baseline and Week 4 of the Maintenance Period (Study Week 17)
Population: Intent to Treat (ITT) Population: all randomized subjects who received at least one dose of study medication, had a Baseline efficacy assessment for the specific outcome, and had at least one respective efficacy outcome assessment collected after randomization (Baseline) visit, i.e. had at least one respective Post-Baseline efficacy assessment.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Treatment Group A: Placebo | Treatment Group B: 2 mg/Day | Treatment Group C: 4 mg/Day | Treatment Group D: 8 mg/Day | Treatment Group E: 12 mg/Day | Treatment Group F: 24 mg/Day
Number analyzed (Participants) | 33 | 13 | 34 | 33 | 34 | 10
Score on a scale | -1.91 [-4.15 to 0.34] | -1.58 [-5.02 to 1.86] | -2.76 [-5.04 to -0.49] | -4.31 [-6.48 to -2.15] | -4.07 [-6.32 to -1.82] | -2.83 [-6.61 to 0.95]
Statistical Analysis 1: Comparison: Treatment Group A: Placebo vs Treatment Group B: 2 mg/Day; Test type: Superiority or Other; p = 0.864, Mixed Models Analysis — P-values are from a Mixed Model Repeated Measures analysis; Mean Difference (Final Values) = 0.33, 95% CI 2-sided [-3.41 to 4.05]
Statistical Analysis 2: Comparison: Treatment Group A: Placebo vs Treatment Group C: 4 mg/Day; Test type: Superiority or Other; p = 0.539, Mixed Models Analysis — P-values are from a Mixed Model Repeated Measures analysis; Mean Difference (Final Values) = -0.85, 95% CI 2-sided [-3.61 to 1.90]
Statistical Analysis 3: Comparison: Treatment Group A: Placebo vs Treatment Group D: 8 mg/Day; Test type: Superiority or Other; p = 0.091, Mixed Models Analysis — P-values are from a Mixed Model Repeated Measures analysis; Mean Difference (Final Values) = -2.40, 95% CI 2-sided [-5.21 to 0.39]
Statistical Analysis 4: Comparison: Treatment Group A: Placebo vs Treatment Group E: 12 mg/Day; Test type: Superiority or Other; p = 0.124, Mixed Models Analysis — P-values are from a Mixed Model Repeated Measures analysis; Mean Difference (Final Values) = -2.16, 95% CI 2-sided [-4.93 to 0.60]
Statistical Analysis 5: Comparison: Treatment Group A: Placebo vs Treatment Group F: 24 mg/Day; Test type: Superiority or Other; p = 0.658, Mixed Models Analysis — P-values are from a Mixed Model Repeated Measures analysis; Mean Difference (Final Values) = -0.92, 95% CI 2-sided [-5.04 to 3.19]
Statistical Analysis 6: Comparison: Treatment Group A: Placebo vs Treatment Group B: 2 mg/Day; Test type: Superiority or Other; p = 0.439, ANCOVA — P-values are from nonparametric rank ANCOVA without stratifications
Statistical Analysis 7: Comparison: Treatment Group A: Placebo vs Treatment Group C: 4 mg/Day; Test type: Superiority or Other; p = 0.177, ANCOVA — P-values are from nonparametric rank ANCOVA without stratifications
Statistical Analysis 8: Comparison: Treatment Group A: Placebo vs Treatment Group D: 8 mg/Day; Test type: Superiority or Other; p = 0.060, ANCOVA — P-values are from nonparametric rank ANCOVA without stratifications
Statistical Analysis 9: Comparison: Treatment Group A: Placebo vs Treatment Group E: 12 mg/Day; Test type: Superiority or Other; p = 0.047, ANCOVA — P-values are from nonparametric rank ANCOVA without stratifications
Statistical Analysis 10: Comparison: Treatment Group A: Placebo vs Treatment Group F: 24 mg/Day; Test type: Superiority or Other; p = 0.407, ANCOVA — P-values are from nonparametric rank ANCOVA without stratifications

2. Secondary Outcome: Number of Participants With a >=5 Points Reduction From Baseline in UPDRS Motor Score
Description: The UPDRS motor scores can range from 0-108 where the maximum score indicates the worse condition. Baseline is defined as the last non-missing assessment measured on or before the first dose date. The change from Baseline will be calculated by subtracting the Baseline values from the individual post-randomization values.
Time Frame: Baseline and Week 4 of the Maintenance Period (Study Week 17)
Population: ITT Population. All participants with a non-missing efficacy observation at Baseline and during the maintenance period were analyzed
Measure: Number; unit: Participants
Arm/Group | Treatment Group A: Placebo | Treatment Group B: 2 mg/Day | Treatment Group C: 4 mg/Day | Treatment Group D: 8 mg/Day | Treatment Group E: 12 mg/Day | Treatment Group F: 24 mg/Day
Number analyzed (Participants) | 35 | 13 | 35 | 33 | 34 | 10
Participants | 9 | 6 | 14 | 16 | 19 | 5
Statistical Analysis 1: Comparison: Treatment Group A: Placebo vs Treatment Group B: 2 mg/Day; Test type: Superiority or Other; p = 0.397, Generalized Estimating Equations model; Odds Ratio (OR) = 2.003, 95% CI 2-sided [0.40 to 9.98]
Statistical Analysis 2: Comparison: Treatment Group A: Placebo vs Treatment Group C: 4 mg/Day; Test type: Superiority or Other; p = 0.131, Generalized Estimating Equations model; Odds Ratio (OR) = 2.242, 95% CI 2-sided [0.79 to 6.40]
Statistical Analysis 3: Comparison: Treatment Group A: Placebo vs Treatment Group D: 8 mg/Day; Test type: Superiority or Other; p = 0.018, Generalized Estimating Equations model; Odds Ratio (OR) = 3.515, 95% CI 2-sided [1.25 to 9.92]
Statistical Analysis 4: Comparison: Treatment Group A: Placebo vs Treatment Group E: 12 mg/Day; Test type: Superiority or Other; p = 0.020, Generalized Estimating Equations model; Odds Ratio (OR) = 3.607, 95% CI [1.22 to 10.64]
Statistical Analysis 5: Comparison: Treatment Group A: Placebo vs Treatment Group F: 24 mg/Day; Test type: Superiority or Other; p = 0.202, Generalized Estimating Equations model; Odds Ratio (OR) = 2.679, 95% CI 2-sided [0.59 to 12.16]

3. Secondary Outcome: Number of Participants With a >=10 Points Reduction From Baseline in UPDRS Motor Score
Description: as for outcome 2
Time Frame: Baseline and Week 4 of the Maintenance Period (Study Week 17)
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Treatment Group A: Placebo | Treatment Group B: 2 mg/Day | Treatment Group C: 4 mg/Day | Treatment Group D: 8 mg/Day | Treatment Group E: 12 mg/Day | Treatment Group F: 24 mg/Day
Number analyzed (Participants) | 35 | 13 | 35 | 33 | 34 | 10
Participants | 5 | 3 | 7 | 7 | 9 | 2
Statistical Analysis 1: Comparison: Treatment Group A: Placebo vs Treatment Group B: 2 mg/Day; Test type: Superiority or Other; p = 0.662, Generalized Estimating Equations model; Odds Ratio (OR) = 1.544, 95% CI [0.22 to 10.84]
Statistical Analysis 2: Comparison: Treatment Group A: Placebo vs Treatment Group C: 4 mg/Day; Test type: Superiority or Other; p = 0.557, Generalized Estimating Equations model; Odds Ratio (OR) = 1.485, 95% CI 2-sided [0.40 to 5.55]
Statistical Analysis 3: Comparison: Treatment Group A: Placebo vs Treatment Group D: 8 mg/Day; Test type: Superiority or Other; p = 0.347, Generalized Estimating Equations model; Odds Ratio (OR) = 1.855, 95% CI 2-sided [0.51 to 6.72]
Statistical Analysis 4: Comparison: Treatment Group A: Placebo vs Treatment Group E: 12 mg/Day; Test type: Superiority or Other; p = 0.379, Generalized Estimating Equations model; Odds Ratio (OR) = 1.776, 95% CI 2-sided [0.49 to 6.38]
Statistical Analysis 5: Comparison: Treatment Group A: Placebo vs Treatment Group F: 24 mg/Day; Test type: Superiority or Other; p = 0.851, Generalized Estimating Equations model; Odds Ratio (OR) = 1.194, 95% CI 2-sided [0.19 to 7.63]

4. Secondary Outcome: Number of Participants With a >=10 Points Reduction From Baseline in UPDRS Parts II and III Combined
Description: The UPDRS Part II is the Activities of Daily Living (ADL) score and can range from 0-52 as determined by the physician. The UPDRS Part III is the Motor Examination (Total Motor Score [TMS]) and is defined as the total score, ranging from 0-108 as determined by the physician, of the tests given in the motor examination section. The combined scores of Parts II and III can range from 0-160 with the higher score indicating the worse condition. Tests were performed when the participant is in the "on" state of Parkinson's. Baseline is defined as the last non-missing assessment measured on or before the first dose date.
Time Frame: Baseline and Week 4 of the Maintenance Period (Study Week 17)
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Treatment Group A: Placebo | Treatment Group B: 2 mg/Day | Treatment Group C: 4 mg/Day | Treatment Group D: 8 mg/Day | Treatment Group E: 12 mg/Day | Treatment Group F: 24 mg/Day
Number analyzed (Participants) | 35 | 13 | 35 | 33 | 34 | 10
Participants | 6 | 3 | 7 | 10 | 12 | 5

5. Secondary Outcome: Responder Rate Defined as Participants With a >=30% Reduction in Baseline UPDRS Motor Score
Description: The responder rate is defined as the percentage of participants with a greater than or equal to (>=)30% reduction in their individual Baseline UPDRS motor score at Week 4 of the Maintenance Period (Study Week 17). Baseline is defined as the last non-missing assessment measured on or before the first dose date. The change from Baseline will be calculated by subtracting the Baseline values from the individual post-randomization values.
Time Frame: Baseline and Week 4 of the Maintenance Period (Study Week 17)
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Treatment Group A: Placebo | Treatment Group B: 2 mg/Day | Treatment Group C: 4 mg/Day | Treatment Group D: 8 mg/Day | Treatment Group E: 12 mg/Day | Treatment Group F: 24 mg/Day
Number analyzed (Participants) | 35 | 13 | 35 | 33 | 34 | 10
Percentage of Participants | 18 | 31 | 23 | 30 | 38 | 31
Statistical Analysis 1: Comparison: Treatment Group A: Placebo vs Treatment Group B: 2 mg/Day; Test type: Superiority or Other; p = 0.540, Generalized Estimating Equations model; Odds Ratio (OR) = 1.591, 95% CI 2-sided [0.36 to 7.03]
Statistical Analysis 2: Comparison: Treatment Group A: Placebo vs Treatment Group C: 4 mg/Day; Test type: Superiority or Other; p = 0.494, Generalized Estimating Equations model; Odds Ratio (OR) = 1.473, 95% CI 2-sided [0.49 to 4.47]
Statistical Analysis 3: Comparison: Treatment Group A: Placebo vs Treatment Group D: 8 mg/Day; Test type: Superiority or Other; p = 0.115, Generalized Estimating Equations model; Odds Ratio (OR) = 2.391, 95% CI 2-sided [0.81 to 7.06]
Statistical Analysis 4: Comparison: Treatment Group A: Placebo vs Treatment Group E: 12 mg/Day; Test type: Superiority or Other; p = 0.045, Generalized Estimating Equations model; Odds Ratio (OR) = 2.960, 95% CI 2-sided [1.02 to 8.55]
Statistical Analysis 5: Comparison: Treatment Group A: Placebo vs Treatment Group F: 24 mg/Day; Test type: Superiority or Other; p = 0.221, Generalized Estimating Equations model; Odds Ratio (OR) = 2.506, 95% CI 2-sided [0.58 to 10.90]

6. Secondary Outcome: Change From Baseline in UPDRS Parts II and III Combined
Description: The UPDRS Part II is the Activities of Daily Living (ADL) score and can range from 0-52 as determined by the physician. The UPDRS Part III is the Motor Examination (Total Motor Score [TMS]) and is defined as the total score, ranging from 0-108 as determined by the physician, of the tests given in the motor examination section. The combined scores of Parts II and III can range from 0-160 with the higher score indicating the worse condition. Tests were performed when the participant is in the "on" state of Parkinson's. Baseline is defined as the last non-missing assessment measured on or before the first dose date. The change from Baseline will be calculated by subtracting the Baseline values from the individual post-randomization values.
Time Frame: Baseline and Week 4 of the Maintenance Period (Study Week 17)
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Treatment Group A: Placebo | Treatment Group B: 2 mg/Day | Treatment Group C: 4 mg/Day | Treatment Group D: 8 mg/Day | Treatment Group E: 12 mg/Day | Treatment Group F: 24 mg/Day
Number analyzed (Participants) | 28 | 13 | 32 | 31 | 32 | 10
Scores on a scale | -2.88 [-5.87 to 0.10] | -1.81 [-6.18 to 2.57] | -3.81 [-6.76 to -0.85] | -5.63 [-8.44 to -2.81] | -6.62 [-9.51 to -3.72] | -3.87 [-8.68 to 0.94]
Statistical Analysis 1: Comparison: Treatment Group A: Placebo vs Treatment Group B: 2 mg/Day; Test type: Superiority or Other; p = 0.662, Mixed Models Analysis — P-values are from a Mixed Model Repeated Measures analysis; Mean Difference (Final Values) = 1.07, 95% CI 2-sided [-3.78 to 5.93]
Statistical Analysis 2: Comparison: Treatment Group A: Placebo vs Treatment Group C: 4 mg/Day; Test type: Superiority or Other; p = 0.621, Mixed Models Analysis — P-values are from a Mixed Model Repeated Measures analysis; Mean Difference (Final Values) = -0.93, 95% CI 2-sided [-4.63 to 2.77]
Statistical Analysis 3: Comparison: Treatment Group A: Placebo vs Treatment Group D: 8 mg/Day; Test type: Superiority or Other; p = 0.150, Mixed Models Analysis — P-values are from a Mixed Model Repeated Measures analysis; Mean Difference (Final Values) = -2.75, 95% CI 2-sided [-6.50 to 1.01]
Statistical Analysis 4: Comparison: Treatment Group A: Placebo vs Treatment Group E: 12 mg/Day; Test type: Superiority or Other; p = 0.048, Mixed Models Analysis — P-values are from a Mixed Model Repeated Measures analysis; Mean Difference (Final Values) = -3.74, 95% CI 2-sided [-7.43 to -0.04]
Statistical Analysis 5: Comparison: Treatment Group A: Placebo vs Treatment Group F: 24 mg/Day; Test type: Superiority or Other; p = 0.715, Mixed Models Analysis — P-values are from a Mixed Model Repeated Measures analysis; Mean Difference (Final Values) = -0.99, 95% CI 2-sided [-6.32 to 4.35]

7. Secondary Outcome: Change From Baseline in UPDRS Activities of Daily Living
Description: The UPDRS Part II is the Activities of Daily Living (ADL) score and can range from 0-52 as determined by the physician. The higher score indicates the worse condition. Tests were performed when the participant is in the "on" state of Parkinson's. Baseline is defined as the last non-missing assessment measured on or before the first dose date. The change from Baseline will be calculated by subtracting the Baseline values from the individual post-randomization values.
Time Frame: Baseline and Week 4 of the Maintenance Period (Study Week 17)
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Treatment Group A: Placebo | Treatment Group B: 2 mg/Day | Treatment Group C: 4 mg/Day | Treatment Group D: 8 mg/Day | Treatment Group E: 12 mg/Day | Treatment Group F: 24 mg/Day
Number analyzed (Participants) | 27 | 11 | 28 | 28 | 25 | 7
Score on a scale | -0.26 [-1.23 to 0.72] | 0.91 [-0.58 to 2.41] | -0.73 [-1.74 to 0.27] | -1.13 [-2.08 to -0.17] | -1.27 [-2.32 to -0.22] | -0.99 [-2.77 to 0.79]
Statistical Analysis 1: Comparison: Treatment Group A: Placebo vs Treatment Group B: 2 mg/Day; Test type: Superiority or Other; p = 0.158, Mixed Models Analysis — P-values are from a Mixed Model Repeated Measures analysis; Mean Difference (Final Values) = 1.17, 95% CI 2-sided [-0.46 to 2.81]
Statistical Analysis 2: Comparison: Treatment Group A: Placebo vs Treatment Group C: 4 mg/Day; Test type: Superiority or Other; p = 0.446, Mixed Models Analysis — P-values are from a Mixed Model Repeated Measures analysis; Mean Difference (Final Values) = -0.47, 95% CI 2-sided [-1.71 to 0.76]
Statistical Analysis 3: Comparison: Treatment Group A: Placebo vs Treatment Group D: 8 mg/Day; Test type: Superiority or Other; p = 0.163, Mixed Models Analysis — P-values are from a Mixed Model Repeated Measures analysis; Mean Difference (Final Values) = -0.87, 95% CI 2-sided [-2.10 to 0.36]
Statistical Analysis 4: Comparison: Treatment Group A: Placebo vs Treatment Group E: 12 mg/Day; Test type: Superiority or Other; p = 0.117, Mixed Models Analysis — P-values are from a Mixed Model Repeated Measures analysis; Mean Difference (Final Values) = -1.01, 95% CI 2-sided [-2.27 to 0.25]
Statistical Analysis 5: Comparison: Treatment Group A: Placebo vs Treatment Group F: 24 mg/Day; Test type: Superiority or Other; p = 0.456, Mixed Models Analysis — P-values are from a Mixed Model Repeated Measures analysis; Mean Difference (Final Values) = -0.73, 95% CI 2-sided [-2.67 to 1.20]

8. Secondary Outcome: Change From Baseline in the Total UPDRS Score (Parts I-III)
Description: The total UPDRS score was calculated by the sum of the values for each component (Part I + Part II + Part III) as determined by the physician. The UPDRS Part I scores mentation, behavior and mood and scores can range from 0-16. The UPDRS Part II is the Activities of Daily Living (ADL) score and can range from 0-52. The UPDRS Part III is the Motor Examination (Total Motor Score [TMS]) and scores range from 0-108. The total UPDRS (Part I + II + III) scores can range from 0-176 with the higher score indicating the worse condition. Tests were performed when the participant is in the "on" state of Parkinson's. Baseline is defined as the last non-missing assessment measured on or before the first dose date. The change from Baseline will be calculated by subtracting the Baseline values from the individual post-randomization values.
Time Frame: Baseline and Week 4 of the Maintenance Period (Study Week 17)
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Treatment Group A: Placebo | Treatment Group B: 2 mg/Day | Treatment Group C: 4 mg/Day | Treatment Group D: 8 mg/Day | Treatment Group E: 12 mg/Day | Treatment Group F: 24 mg/Day
Number analyzed (Participants) | 28 | 13 | 32 | 31 | 32 | 10
Score on a scale | -2.74 [-5.79 to 0.31] | -2.18 [-6.65 to 2.29] | -3.83 [-6.85 to -0.81] | -5.93 [-8.80 to -3.06] | -6.68 [-9.64 to -3.71] | -3.40 [-8.30 to 1.50]
Statistical Analysis 1: Comparison: Treatment Group A: Placebo vs Treatment Group B: 2 mg/Day; Test type: Superiority or Other; p = 0.823, Mixed Models Analysis — P-values are from a Mixed Model Repeated Measures analysis; Mean Difference (Final Values) = 0.56, 95% CI 2-sided [-4.38 to 5.50]
Statistical Analysis 2: Comparison: Treatment Group A: Placebo vs Treatment Group C: 4 mg/Day; Test type: Superiority or Other; p = 0.568, Mixed Models Analysis — P-values are from a Mixed Model Repeated Measures analysis; Mean Difference (Final Values) = -1.09, 95% CI 2-sided [-4.86 to 2.68]
Statistical Analysis 3: Comparison: Treatment Group A: Placebo vs Treatment Group D: 8 mg/Day; Test type: Superiority or Other; p = 0.101, Mixed Models Analysis — P-values are from a Mixed Model Repeated Measures analysis; Mean Difference (Final Values) = -3.19, 95% CI 2-sided [-7.01 to 0.63]
Statistical Analysis 4: Comparison: Treatment Group A: Placebo vs Treatment Group E: 12 mg/Day; Test type: Superiority or Other; p = 0.040, Mixed Models Analysis — P-values are from a Mixed Model Repeated Measures analysis; Mean Difference (Final Values) = -3.94, 95% CI 2-sided [-7.70 to -0.18]
Statistical Analysis 5: Comparison: Treatment Group A: Placebo vs Treatment Group F: 24 mg/Day; Test type: Superiority or Other; p = 0.811, Mixed Models Analysis — P-values are from a Mixed Model Repeated Measures analysis; Mean Difference (Final Values) = -0.66, 95% CI 2-sided [-6.08 to 4.77]

9. Secondary Outcome: Change From Baseline in the UPDRS Part I (Mentation)
Description: The UPDRS Part I scores mentation, behavior and mood as determined by a physician and participants were tested during the "on" phase of Parkinson's. This component of the UPDRS is the total score for 4 items (the items 1- 4 include intellectual impairment, thought disorder, motivation/initiative, and depression) and may have a value ranging from 0 to 16 as determined by a physician where 16 indicates the maximum score and the worse condition. All 4 items have to be present for a total score to be calculated. If one or more items are missing, the total score for the component will also be missing. Baseline is defined as the last non-missing assessment measured on or before the first dose date. The change from Baseline will be calculated by subtracting the Baseline values from the individual post-randomization values.
Time Frame: Baseline and Week 4 of the Maintenance Period (Study Week 17)
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Treatment Group A: Placebo | Treatment Group B: 2 mg/Day | Treatment Group C: 4 mg/Day | Treatment Group D: 8 mg/Day | Treatment Group E: 12 mg/Day | Treatment Group F: 24 mg/Day
Number analyzed (Participants) | 33 | 13 | 34 | 33 | 34 | 10
Score on a scale | 0.05 [-0.24 to 0.34] | -0.34 [-0.78 to 0.10] | -0.01 [-0.31 to 0.28] | -0.26 [-0.54 to 0.02] | -0.02 [-0.31 to 0.27] | 0.50 [0.02 to 0.98]
Statistical Analysis 1: Comparison: Treatment Group A: Placebo vs Treatment Group B: 2 mg/Day; Test type: Superiority or Other; p = 0.102, Mixed Models Analysis — P-values are from a Mixed Model Repeated Measures analysis; Mean Difference (Final Values) = -0.39, 95% CI 2-sided [-0.86 to 0.08]
Statistical Analysis 2: Comparison: Treatment Group A: Placebo vs Treatment Group C: 4 mg/Day; Test type: Superiority or Other; p = 0.723, Mixed Models Analysis — P-values are from a Mixed Model Repeated Measures analysis; Mean Difference (Final Values) = -0.06, 95% CI 2-sided [-0.41 to 0.29]
Statistical Analysis 3: Comparison: Treatment Group A: Placebo vs Treatment Group D: 8 mg/Day; Test type: Superiority or Other; p = 0.084, Mixed Models Analysis — P-values are from a Mixed Model Repeated Measures analysis; Mean Difference (Final Values) = -0.31, 95% CI 2-sided [-0.66 to 0.04]
Statistical Analysis 4: Comparison: Treatment Group A: Placebo vs Treatment Group E: 12 mg/Day; Test type: Superiority or Other; p = 0.697, Mixed Models Analysis — P-values are from a Mixed Model Repeated Measures analysis; Mean Difference (Final Values) = -0.07, 95% CI 2-sided [-0.42 to 0.28]
Statistical Analysis 5: Comparison: Treatment Group A: Placebo vs Treatment Group F: 24 mg/Day; Test type: Superiority or Other; p = 0.086, Mixed Models Analysis — P-values are from a Mixed Model Repeated Measures analysis; Mean Difference (Final Values) = 0.45, 95% CI 2-sided [-0.06 to 0.97]

10. Secondary Outcome: Responder Rate According to the Clinical Global Impression - Global Improvement (CGI-I) Scale
Description: The CGI-I scale allows the investigator to rate the participant's total improvement since the beginning of treatment (Baseline). Baseline is defined as the last non-missing assessment measured on or before the first dose date. The scale is rated from 1-7 where 1 = "very much improved", 2 = "much improved", 3 = "minimally improved", 4 = "no change", 5 = "minimally worse, 6 = "much worse", and 7 = "very much worse". The responder rate is defined as the percentage of participants with a score of 1 or 2.
Time Frame: Week 4 of the Maintenance Period (Study Week 17)
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Treatment Group A: Placebo | Treatment Group B: 2 mg/Day | Treatment Group C: 4 mg/Day | Treatment Group D: 8 mg/Day | Treatment Group E: 12 mg/Day | Treatment Group F: 24 mg/Day
Number analyzed (Participants) | 40 | 13 | 40 | 40 | 39 | 13
Percentage of participants | 20 | 15 | 28 | 45 | 56 | 23
Statistical Analysis 1: Comparison: Treatment Group A: Placebo vs Treatment Group B: 2 mg/Day; Test type: Superiority or Other; p = 0.733, Generalized Estimating Equations model; Odds Ratio (OR) = 0.769, 95% CI 2-sided [0.17 to 3.49]
Statistical Analysis 2: Comparison: Treatment Group A: Placebo vs Treatment Group C: 4 mg/Day; Test type: Superiority or Other; p = 0.519, Generalized Estimating Equations model; Odds Ratio (OR) = 1.411, 95% CI 2-sided [0.50 to 4.02]
Statistical Analysis 3: Comparison: Treatment Group A: Placebo vs Treatment Group D: 8 mg/Day; Test type: Superiority or Other; p = 0.008, Generalized Estimating Equations model; Odds Ratio (OR) = 4.204, 95% CI 2-sided [1.46 to 12.07]
Statistical Analysis 4: Comparison: Treatment Group A: Placebo vs Treatment Group E: 12 mg/Day; Test type: Superiority or Other; p = 0.001, Generalized Estimating Equations model; Odds Ratio (OR) = 5.456, 95% CI 2-sided [1.93 to 15.46]
Statistical Analysis 5: Comparison: Treatment Group A: Placebo vs Treatment Group F: 24 mg/Day; Test type: Superiority or Other; p = 0.752, Generalized Estimating Equations model; Odds Ratio (OR) = 1.281, 95% CI 2-sided [0.27 to 5.98]

11. Secondary Outcome: Percentage of Participants Withdrawn From the Study Due to Lack of Efficacy
Description: The percentage of participants who withdrew from the study due to lack of efficacy as defined by either the participant or the investigator is presented here.
Time Frame: Up to Week 4 of the Maintenance Period (Study Week 17)
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Treatment Group A: Placebo | Treatment Group B: 2 mg/Day | Treatment Group C: 4 mg/Day | Treatment Group D: 8 mg/Day | Treatment Group E: 12 mg/Day | Treatment Group F: 24 mg/Day
Number analyzed (Participants) | 40 | 13 | 40 | 40 | 39 | 13
Percentage of participants | 5 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious AEs were collected from the initial dose of study treatment through the completion of the Follow-up Period (up to 28 weeks)
Description: An AE is any untoward medical occurrence in a participant temporally associated with the use of a medicinal product, whether or not considered related to the study treatment. A SAE results in death, is life-threatening, requires hospitalization, results in disability or incapacity, or is a congenital anomaly or birth defect.
Arm/Group | Treatment Group A: Placebo | Treatment Group B: 2 mg/Day | Treatment Group C: 4 mg/Day | Treatment Group D: 8 mg/Day | Treatment Group E: 12 mg/Day | Treatment Group F: 24 mg/Day
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/13 | 1/41 | 0/40 | 2/39 | 0/13
Other Adverse Events (participants affected / at risk) | 17/40 | 5/13 | 18/41 | 24/40 | 18/39 | 7/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Group A: Placebo (N=40) | Treatment Group B: 2 mg/Day (N=13) | Treatment Group C: 4 mg/Day (N=41) | Treatment Group D: 8 mg/Day (N=40) | Treatment Group E: 12 mg/Day (N=39) | Treatment Group F: 24 mg/Day (N=13)
Cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Group A: Placebo (N=40) | Treatment Group B: 2 mg/Day (N=13) | Treatment Group C: 4 mg/Day (N=41) | Treatment Group D: 8 mg/Day (N=40) | Treatment Group E: 12 mg/Day (N=39) | Treatment Group F: 24 mg/Day (N=13)
Somnolence (Nervous system disorders) | 2 | 2 | 5 | 4 | 3 | 1
Headache (Nervous system disorders) | 1 | 1 | 4 | 3 | 2 | 2
Dizziness (Nervous system disorders) | 2 | 0 | 2 | 4 | 3 | 1
Sudden onset of sleep (Nervous system disorders) | 0 | 0 | 2 | 0 | 4 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1
Tremor (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1
Dizziness postural (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 3 | 1 | 6 | 13 | 4 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0 | 3 | 3 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 1 | 1 | 3 | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 0 | 2 | 4 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 1 | 0
Nasopharyngitis (Infections and infestations) | 3 | 0 | 1 | 2 | 2 | 0
Pyelonephritis chronic (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 1 | 1 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 2 | 2 | 1 | 2
Labile blood pressure (Vascular disorders) | 0 | 0 | 0 | 1 | 1 | 1
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 2 | 0
Blood creatine (Investigations) | 0 | 0 | 1 | 2 | 1 | 1
Abnormal dreams (Psychiatric disorders) | 2 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Libido increased (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 2 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 3 | 1
Back injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Skeletal injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Dysplastic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.